CLINICAL TRIAL: NCT02683226
Title: Comparison of Alogliptin Versus Alogliptin and Pioglitazone on Insulin Resistance of Metformin Treated Women With PCOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Andrej Janez, Andrej Janez, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTT
Record Dates: First submitted 2016-02-11; First posted 2016-02-17 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2015-02

CONDITIONS: Polycystic Ovary Syndrome; Insulin Resistance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance

ARMS (2):
- metformin and alogliptin (Experimental): Vipdomet 12.5 mg/1000 mg tablets
  Interventions: Drug: Vipdomet
- pioglitasone and alogliptin (Experimental): Incresync 12,5 mg/30 mg tablets
  Interventions: Drug: Incresync

INTERVENTIONS:
Drug: Vipdomet
  Arms: metformin and alogliptin
Drug: Incresync
  Arms: pioglitasone and alogliptin

SUMMARY:
The purpose of this study was to determine whether dual treatment with metformin and alogliptin is more effective than treatment with metformin, alogliptin and pioglitazone in the treatment of obese women with polycystic ovary syndrome (PCOS) regarding insulin resistance and beta cell function.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old to menopause
* polycystic ovary syndrome (NICHD criteria)
* BMI of 30 kg/m² or higher

Exclusion Criteria:

* type 1 or type 2 diabetes mellitus
* history of carcinoma
* Cushing's syndrome or congenital (non-classic) adrenal hyperplasia
* personal or family history of MEN 2
* significant cardiovascular, kidney or hepatic disease

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The main outcome was change in insulin resistance measured with homeostasis model assessment (HOMA IR). | HOMA IR was calculated at the base point and at the endpoint of 12 weeks of clinical trial.
  HOMA IR was calculated as the product of the fasting glucose and insulin concentration divided by 22,5.
Primary outcome was change in beta cell function using adaptation index. | Adaptation index was calculated at the base point and at the endpoint of 12 weeks of clinical trial.
  Adaptation index was calculated using the product between prehepatic insulin delivery and oral glucose insulin sensitivity (OGIS), calculated using online calculator.
Primary outcome was change in fasting concentration of glucose. | Patient's fasting blood was drawn at the base point and at the endpoint of 12 weeks of clinical trial.
  Patient's blood was drawn between 8 and 9 a.m. Concentrations of fasting glucose was measured in mmol/L.
Primary outcome was change in fasting concentration of insulin. | Patient's fasting blood was drawn at the base point and at the endpoint of 12 weeks of clinical trial.
  Patient's blood was drawn between 8 and 9 a.m. Concentrations of fasting insulin was measured in mU/L.

SECONDARY OUTCOMES:
Secondary outcome was change in body mass index (BMI). | Patient's body weight were measured at the base point and every four weeks during the 12 weeks of clinical trial. Patient's height was measured at the basepoint
  Patient's BMI was defined as the patient's body mass in kilograms divided by the square of their height in meters.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia